CLINICAL TRIAL: NCT03953248
Title: L-Carnitine as an Adjuvant Treatment in Acute Phosphide Poisoning (LC): A Randomized Clinical Trial
Brief Title: L-Carnitine as an Adjuvant Treatment in Acute Phosphide Poisoning (LC)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Heba Allah Ali Abd El-Halim Mabrouk (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Heba Allah Ali Abd El-Halim Mabrouk, Principal Investigator, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LC-2018-CT; L-Carnitine (Registry Identifier: LC)
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Toxicity
Keywords: phosphide; poisoning; L-carnitine; oxidative stress
MeSH Terms: conditions — Poisoning | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No

ARMS (2):
- Non L-Carnitine (No Intervention): Subjects in this arm will receive standard treatment only (without LC). It consists of patient resuscitation, gastric decontamination (with sodium bicarbonate, and activated charcoal [1 g/Kg, orally] in the first 6 hours after onset of poisoning), adequate hydration and supportive treatment
- L-Carnitine (Active Comparator): Subjects in this arm will receive standard treatment in addition to LC IV, as a dose of 1 g/8 hours
  Interventions: Drug: L-Carnitine

INTERVENTIONS:
Drug: L-Carnitine
  Arms: L-Carnitine

SUMMARY:
The aim of this study was to evaluate efficacy and safety of Alpha Lipoic Acid(ALA) as an adjuvant in the management of patients with acute phosphide poisoning.

DETAILED DESCRIPTION:
The study was carried out following approval of the research ethical committee of Tanta Faculty of Medicine on patients admitted to The Poison Control Unit (Emergency Hospitals, Tanta and Mansoura Universities) with acute phosphide poisoning in the period from January 2016 to January 2018. A written informed consent was taken from each patient or his/her guardians (if the patient was unable to participate in the consent process). Confidentiality of the data was maintained by making code numbers for each patient. The investigators planned to conduct a randomized clinical trial to evaluate efficacy and safety of LC as an adjuvant in treatment of patients with acute phosphide poisoning. Fifty patients was randomized to LC or a non LC in a 1:1 ratio (25 patients in each group). LC was given IV, as a dose of 1 g/8 hours. Patients was monitored and a detailed documentation of any adverse effect due to LC therapy was recorded.

This intervention represented an added treatment to the existing standard of care. All patients will continue to receive standard treatment, which was determined by the attending physician who maintained clinical responsibility for all patients. It consisted of patient resuscitation, gastric decontamination (with sodium bicarbonate, and activated charcoal [1 g/Kg, orally] in the first 6 hours after onset of poisoning), adequate hydration and supportive treatment. All the patients was followed up until discharge or death. All patients was subjected to:

I. History. II. Clinical examination. III. Laboratory investigations: At admission and repeated before discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female, aged 12 years or older) with symptomatic acute phosphide poisoning (deliberate or accidental), with diagnosis made on the basis of:

The typical clinical manifestations due to and following shortly after a single exposure to phosphide.

Reliable identification of the compound based on the container brought by patient attendants or a subsequent confirmation by silver nitrate test for phosphine detection in stomach contents.

Exclusion Criteria:

* Patients less than 12 years of age Pregnant and lactating women Patients with ingestion or exposure to other substances in addition to phosphide.

Patients with other major medical conditions (e.g. cardiovascular disease, renal or hepatic failure).

Patients presenting more than 6 hours of having consumed the phosphide compound (late presenters).

Patients treated for acute phosphide poisoning in any medical center before admission

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 2 years
  Death Rate

SECONDARY OUTCOMES:
Duration of hospital stay | 2 years
  Duration that patient will stay in hospital

OTHER OUTCOMES:
Need for intubation | 2 years
  will the patient need to be intubated or not

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years